CLINICAL TRIAL: NCT04761419
Title: Effect of Parents' Presence in Nagano Children's Hospital NICU on Infant and Parent Outcomes
Brief Title: Family Centered Care Cohort Study 1 in Nagano Children's Hospital
Status: Active, not recruiting | Type: Observational
Sponsor: Nagano Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FCC-cohort1
Record Dates: First submitted 2021-02-12; First posted 2021-02-18 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Family Centered Care
MeSH Terms: interventions — Infant Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: Parents' longer presence beside their infant — They are not intervention. We will collect data about these items.
  Other Names: Parents' longer skin-to-skin contact; Parents' longer participation in infant care; Parents' longer interaction with their infant

SUMMARY:
An observational cohort study to show the effect of parents' presence beside their infants, skin-to-skin contact (SCC), participation in infant care, or any interaction with their infants on parents' and infants' short- and long-term outcomes. Investigators create a hypothesis that longer parents' presence, SCC, participation in infant care, and any interaction with their infants affect outcomes of infants and parents by preventing parents' depression and promoting parent-infant bonding and, in addition, by shortening the length of stay, promoting growth, promoting establishment breastfeeding, and improving developmental outcomes. Parents are asked to make a record of the length of their presence, SCC, participation in infant care, and any interaction with their infants, which are quantitative measurements of family centered care (FCC). Investigators also collect the data related to the background information of the family, delivery, the clinical course of infants, and the outcome measures of the infants and parents. No intervention is included in this research.

The study setting is a level IV neonatal intensive care unit (NICU) at Nagano Children's Hospital in Nagano, Japan. Eligible infants are those who are born at 34 weeks of gestation or earlier from Japanese parents in Nagano Children's Hospital and need admission into NICU in the same hospital. Infants are excluded from this study if they have any major anomalies including suspicion of chromosomal disorder on admission, if at least one parent is Not Japanese, or if they do not survive until discharge home.

The primary outcomes are the EPDS and Japanese version of Mother-to-Infant Bonding Scale (MIBS-J) of the parents. The secondary outcomes are the followings; (1) length of stay (days), (2) physical measurements at 36 weeks (g or cm) and growth rate from birth to discharge home (g or cm /d), (3) breastmilk-feeding (exclusive, partial, or no breast milk) and the frequency of breastfeeding directly from breast at 36 weeks PMA and at discharge (average frequency per day), and for the infants whose birth weight <1500g only, (4) developmental quotient (DQ) at 6 and 18 months of corrected age, and 3 years old assessed by Kyoto Scale of Psychological Development (KSPD).

DETAILED DESCRIPTION:
<Ethical considerations> This research protocol was approved by the Ethics Committee of Nagano Children's Hospital before this research is being conducted. Recruitment is undertaken by the neonatologists in the unit. They provide written and oral information about the study when they explain infants' condition to their parents at admission. The parents are given sufficient time to consider their participation. The informed consent will be asked within 7 days from the birth, otherwise the infant will be excluded from this study. At least one of the parents should sign the informed consent before enrolment. At the time of agreement, investigators give the infant an anonymous number to protect personal information.

< Power calculation > The sample size should be decided by the number of parents as the primary outcomes are for parents. Investigators plan to include 110 couples or families; the power calculation showed that investigators could detect a 2.5 difference in the mean Edinburgh Postnatal Depression Scale (EPDS) score of longer and shorter presence groups (with power 0.8 and alfa 0.05) with this number of parents.

<Measures and data collection> Diary record Parents make a record on daily diary from the next day of agreement to one day before discharge. Parents make a record about duration of these four topics; presence, skin-to-skin contact (SCC), participation in infant care, and any other interaction with their infants.

* "Care taking" includes the followings; breast feeding, bottle feeding, milking, tube feeding, changing diaper, wiping body, bathing, and any other essential care for baby. However, any care taking during "SCC" mustn't included in this section.
* "Other interaction with baby" includes the followings; hugging, holding, touching, watching, talking, reading books, playing, making something or writing diary for baby, and any other approaches for baby. However, any interaction given during "SCC" or "care taking" mustn't included in this section.

Investigators use the modified Parent-Infant Closeness Diary. The original diary includes three items for each mother and father; presence, holding and SCC. Investigators have changed these items into our own settings as above and changed the used language into Japanese. Investigators already have got the permission from the developers of this diary. This diary has one day per page including all the four topics for both parents. Mother and father respectively draw a line on the blank of specific items they do. They should fill all the corresponding blanks when they do things for multiple babies. The start and the end times should be put in 5-minute increments. The validity of Parent-Infant Closeness Diary has already been proven.

Perinatal Data Collection Perinatal information of the infant includes sex, gestational age, birth weight, height, head circumference, mode of delivery, parity and plurality of mother, and Apgar score at 1, 5, and 10 minutes. Investigators will also find out if the infant meets the criteria for small for gestational age (SGA), which is defined as both birth weight and height are <10th percentile.

Perinatal information of the family members includes the first meeting days with the infant and the first SCC days, for mother and father respectively.

Background information of the family includes family composition, presence of mother's supporter, the number of siblings living with parents, and required time from home to the hospital.

Background information of the parents includes the age, the educational background, the smoking history at pregnant, occupation and parental leave, history of depression or any other mental health problem before and during pregnancy and the history of medication for that disease, and the degree of social support, which is measured by the Multidimensional Scale of Perceived Social Support (MSPSS) as mentioned below. These are risk factors of postpartum depression.

Short version of Multidimensional Scale of Perceived Social Support in Japanese (MSPSS-Js) The Multidimensional Scale of Perceived Social Support (MSPSS) is widely used self-report measure of subjectively assessed social support. There have been several modifications for MSPSS and now it consists of 12 questions with 7-point rating scale ranging from very strongly disagree (1) to very strongly agree (7) for each question. There is Japanese version of MSPSS (MSPSS-J), whose reliability and validity have proven. Investigators use short version of MSPSS-J (MSPSS-Js), which consists of only 7 questions with 7-point rating scale ranging from 1 to 7 and has high correlation with full version. The total score varies from minimum 7 to maximum 49, and higher scores indicates to have better social support.

Data Collection of the clinical course The information of the clinical course includes days of invasive ventilation, days of non-invasive ventilation, days of any respiratory support including oxygen, the history of patent ductus arteriosus (PDA) operation, the history of surgical treatment of abdomen, age of full feeding (the amount of enteral nutrition >=100ml/kg/day), the history and the degree of intraventricular hemorrhage (IVH), and the history of retinopathy of prematurity (ROP) treatment.

Evaluation at 36 weeks postmenstrual age (PMA) and discharge Investigators measure the weight (g), height (cm), head circumference(cm), the frequency of breast feeding (per day), and the type of nutrition (exclusive, partial, or no breast milk) at 36 weeks PMA and when the infant discharges home or leaves our NICU to another hospital or ward to prepare for discharge. Investigators also calculate the length of hospital stay (days) and the growth rate of physical measurements between the time of admission and discharge. If the infant leaves our NICU before 36 weeks PMA, investigators use the data at that point as an evaluation at 36 weeks PMA.

The Edinburgh Postnatal Depression Scale (EPDS) and Japanese version of Mother-to-Infant Bonding Scale (MIBS-J) for mother and father All mothers and fathers of the infants enrolled in this research undergo the Edinburgh Postnatal Depression Scale (EPDS) and Japanese version of Mother-to-Infant Bonding Scale (MIBS-J) at least twice. Almost all mothers who deliver in Nagano Children's Hospital usually undergo the EPDS and MIBS-J at 2 and 4 weeks postpartum at the maternity outpatient clinic. Investigators additionally carry out the EPDS and MIBS-J for fathers in NICU once within a month postpartum, and for both fathers and mothers at discharge of their infant for the purpose of this research.

The EPDS is a screening method for mothers to detect postpartum depressive symptoms. It comprises 10 self-report items, each of which is scored on a four-point scale (0-3). The total score varies from minimum 0 to maximum 30, and higher scores indicates to have more depressive symptoms. Investigators use Japanese version of the EPDS, whose reliability and validity have already proven. The cutoff score for Japanese people to indicate probable major postpartum depression should be eight and nine, which is lower than that usually used in western countries.

Mother-to-Infant Bonding Scale (MIBS) is an assessment method for the feelings of a mother towards her new infant, but investigators use Japanese version of MIBS (MIBS-J), whose reliability and validity have already proven. MIBS comprises eight self-report items, but MIBS-J have ten self-report items, each of which is scored on a four-point scale (0-3). The total score varies from minimum 0 to maximum 30, and higher scores indicate a problematic bonding between a mother and her infant.

The main risk factors of mothers' postpartum depression are prenatal depression and anxiety, previous depression or other mental problems, lower income and occupational status, multiparity, presence of other children, poor marital relationship or without partner, lack of social support, stressful life events, negative image toward pregnancy, and experiences of early mother-infant separation. In addition, the risk factors vary depending on when to evaluate postpartum depression. The depression scores in mothers and fathers of preterm infants is at its highest just after delivery and will reduce over time, which shows different change compared with term birth. This is why investigators have to adjust these confounding factors when investigators evaluate the EPDS and MIBS-J of the parents.

Long-term developmental assessment after discharge (birth weight <1500g) The development of the infants whose birth weight <1500g are assessed by Kyoto Scale of Psychological Development (KSPD) at 6 and 18 months of corrected age, and 3 years old at the outpatient clinic of Nagano Children's Hospital. KSPD is one of the assessment methods to evaluate developmental quotient and it is known to be well correlated with Bayley III. KSPD consists of three subscales: Cognitive-Adaptive, Language-Social, and Postural-Motor.

<Outcomes> The primary outcomes are the EPDS and Japanese version of Mother-to-Infant Bonding Scale (MIBS-J) of the parents. Investigators hypothesize that longer parents' presence decreases the EPDS score and MIBS-J score. Investigators will divide mothers and fathers into two groups respectively (longer and shorter presence groups) based on the distribution of the time of parents' presence, and compare the difference of the mean EPDS score and MIBS-J score between these two groups at each point in time measured.

The secondary outcomes are the followings; (1) length of stay (days), (2) physical measurements at 36 weeks (g or cm) and growth rate from birth to discharge home (g or cm /d), (3) breastmilk-feeding (exclusive, partial, or no breast milk) and the frequency of breastfeeding directly from breast at 36 weeks PMA and at discharge (average frequency per day), and for the infants whose birth weight <1500g only, (4) developmental quotient (DQ) at 6 and 18 months of corrected age, and 3 years old assessed by KSPD. Investigators hypothesize that longer parents' presence, SCC, participation in infant care, or any interaction with infant improve these outcomes. Investigators will divide mothers and fathers into two groups respectively (longer and shorter presence groups, SCC, participation in infant care, or any interaction with infant) as mentioned above and compare the difference of these outcomes between these two groups. In addition, investigators also correct the data from the diary as the followings; presence of at least one of their parents, SCC with at least one of their parents, participation of at least one of their parents in infant care, and any interaction with at least one of their parents, and consider the outcomes in the same manner. Investigators will also consider (5) the difference of the mean EPDS score and MIBS-J score between longer and shorter SCC, participation in infant care, or any interaction with infant groups.

<Statistical analysis> As a statistical analysis, investigators will use a mixed effect model for the EPDS score and MIBS-J score, a linear regression model for other continuous variables (length of stay, physical measurements, growth rate, the frequency of breastfeeding and DQ), and a logistic regression model for binary variable (type of nutrition). Potential confounders will be adjusted.

ELIGIBILITY:
Inclusion Criteria:

* Born at 34 weeks of gestation or earlier in Nagano Children's Hospital and need admission into NICU in the same hospital

Exclusion Criteria:

* Having any major anomalies including suspicion of chromosomal disorder on admission
* At least one parent is Not Japanese
* The consent is not obtained by day 7
* Do not survive until discharge home

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A level IV NICU in Japan
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-03-16 (Actual); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
The Edinburgh Postnatal Depression Scale (EPDS) of mother 1 | 2 weeks postpartum.
  Indicators to estimate depression in parents. The total score varies from minimum 0 to maximum 30, and higher scores indicates to have more depressive symptoms.
The Edinburgh Postnatal Depression Scale (EPDS) of mother 2 | 4 weeks postpartum.
  Indicators to estimate depression in parents. The total score varies from minimum 0 to maximum 30, and higher scores indicates to have more depressive symptoms.
The Edinburgh Postnatal Depression Scale (EPDS) of mother 3 | At discharge of the infant, an average of 2 months postpartum.
  Indicators to estimate depression in parents. The total score varies from minimum 0 to maximum 30, and higher scores indicates to have more depressive symptoms.
The Edinburgh Postnatal Depression Scale (EPDS) of father 1 | Within 1 month postpartum.
  Indicators to estimate depression in parents. The total score varies from minimum 0 to maximum 30, and higher scores indicates to have more depressive symptoms.
The Edinburgh Postnatal Depression Scale (EPDS) of father 2 | At discharge of the infant, an average of 2 months postpartum.
  Indicators to estimate depression in parents. The total score varies from minimum 0 to maximum 30, and higher scores indicates to have more depressive symptoms.
Japanese version of Mother-to-Infant Bonding Scale (MIBS-J) for mother 1 | 2 weeks postpartum.
  Indicators to estimate bonding between infant and parents. The total score varies from minimum 0 to maximum 30, and higher scores indicate a problematic bonding between a mother and her infant.
Japanese version of Mother-to-Infant Bonding Scale (MIBS-J) for mother 2 | 4 weeks postpartum.
  Indicators to estimate bonding between infant and parents. The total score varies from minimum 0 to maximum 30, and higher scores indicate a problematic bonding between a mother and her infant.
Japanese version of Mother-to-Infant Bonding Scale (MIBS-J) for mother 3 | At discharge of the infant, an average of 2 months postpartum.
  Indicators to estimate bonding between infant and parents. The total score varies from minimum 0 to maximum 30, and higher scores indicate a problematic bonding between a mother and her infant.
Japanese version of Mother-to-Infant Bonding Scale (MIBS-J) for father 1 | Within 1 month postpartum.
  Indicators to estimate bonding between infant and parents. The total score varies from minimum 0 to maximum 30, and higher scores indicate a problematic bonding between a mother and her infant.
Japanese version of Mother-to-Infant Bonding Scale (MIBS-J) for father 2 | At discharge of the infant, an average of 2 months postpartum.
  Indicators to estimate bonding between infant and parents. The total score varies from minimum 0 to maximum 30, and higher scores indicate a problematic bonding between a mother and her infant.

SECONDARY OUTCOMES:
Length of stay | At discharge of the infant, an average of 2 months postpartum.
  Hospitalization of the infant in NICU
Weight at 36 weeks | 36 weeks of postmenstrual age.
  Weight in grams.
Height at 36 weeks | 36 weeks of postmenstrual age.
  Height in centimeters.
Head circumference at 36 weeks | 36 weeks of postmenstrual age.
  Head circumference in centimeters.
Growth rate of weight from birth to discharge home (change) | At birth and discharge, an average of 2 months postpartum.
  Weight in grams per day
Growth rate of height from birth to discharge home (change) | At birth and discharge, an average of 2 months postpartum.
  Height in centimeters per day
Growth rate of head circumference from birth to discharge home (change) | At birth and discharge, an average of 2 months postpartum.
  Head circumference in centimeters per day
Breastmilk-feeding at 36 weeks | 36 weeks of postmenstrual age.
  Exclusive, partial, or no breast milk
Breastmilk-feeding at discharge | At discharge, an average of 2 months postpartum.
  Exclusive, partial, or no breast milk
Frequency of breastfeeding directly from breast at 36 weeks | 36 weeks of postmenstrual age.
  Average frequency per day
Frequency of breastfeeding directly from breast at discharge | At discharge, an average of 2 months postpartum.
  Average frequency per day
Developmental quotient (DQ) at 6 months of corrected age | At 6 months of corrected age.
  Assessed by Kyoto Scale of Psychological Development (KSPD), which is calculated by dividing the age of the group into which test scores place the child by the child's corrected age and multiplying by 100. Higher score indicates better development.
Developmental quotient (DQ) at 18 months of corrected age | At 18 months of corrected age.
  Assessed by Kyoto Scale of Psychological Development (KSPD), which is calculated by dividing the age of the group into which test scores place the child by the child's corrected age and multiplying by 100. Higher score indicates better development.
Developmental quotient (DQ) at 3 years old | 3 years old (3 years of postmenstrual age)
  Assessed by Kyoto Scale of Psychological Development (KSPD), which is calculated by dividing the age of the group into which test scores place the child by the child's real age and multiplying by 100. Higher score indicates better development.

CONTACTS AND LOCATIONS:
Overall Officials: Ryo Itoshima, MD, Principal Investigator — Nagano Children's Hospital
Locations (1):
- Nagano Children's Hospital, Azumino, Nagano, Japan

IPD SHARING:
Plan to Share IPD: No